CLINICAL TRIAL: NCT05103436
Title: Electrical Stimulation for Spasticity in Spinal Cord Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00112681
Record Dates: First submitted 2021-10-07; First posted 2021-11-02 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either receive 2 months of TENS (1 hr AM, 1 hr PM/day, 50 Hz, below pain/motor threshold, using a EMS 7500 TENS unit) upon entry to the study (Intervention group) or not (Control; but offered the same TENS following a 2-month delay for equipoise).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Participants will not receive intervention for the first 2 months. This period will be used for comparison with the intervention group. At the end of the 2-month delay, they will receive TENS (1 hr AM, 1 hr PM/day, 50 Hz, below pain/motor threshold, using an EMS 7500 TENS unit).
- Intervention Group (Experimental): Participants will receive 2 months of TENS (1 hr AM, 1 hr PM/day, 50 Hz, below pain/motor threshold, using an EMS 7500 TENS unit) immediately upon entry to the study.
  Interventions: Other: TENS

INTERVENTIONS:
Other: TENS — Electrical nerve stimulation
  Arms: Intervention Group

SUMMARY:
This study examines the immediate and long-term effects of lumbosacral TENS on spasticity and residual voluntary force control in spinal cord injury in comparison to no TENS. Participants in the intervention group will receive 2 months of TENS. Participants in the control group will receive TENS after a 2-month delay. Modified Ashworth score and pendulum test will be used to assess spasticity and force control. Electrophysiological measures will be used to assess the activity profile of motorneurons.

DETAILED DESCRIPTION:
Transcutaneous electrical nerve stimulation (TENS) has been used to control pain in stroke, MS, cerebral palsy and spinal cord injury (SCI) and its effect on spasticity reduction, although not used clinically, has been examined recently. In the few SCI studies done to date, the TENS electrodes have been placed on the nerve to the muscle under study and initial reports show a consistent decrease in spasticity measures, like the Modified Ashworth Score (MAS) and reflexes, during or hours after the TENS application. Recently, study team members from the ReYu Recovery Centre in Edmonton have observed that when TENS is applied with both electrodes over the lower back (lumbosacral TENS), varying amounts of immediate and long-term spasticity relief are produced in both legs.

The investigators have observed 3 clients from ReYU and all have shown immediate reductions in spasticity for at least 2 joints in both legs. The effect of the lumbosacral TENS varied from an immediate dramatic reduction to a more moderate reduction when applied over several days. This study will examine the immediate and longer-term (2 months) effect of using spinal TENS in reducing spasticity of the lower limbs in a larger number of participants with SCI. The investigators want to understand how spinal TENS affects spinal circuits and motoneurons below the lesion to reduce spasticity to observe improvement in its effect in those with more moderate responses. Lumbosacral TENS has the potential for a non-pharmacological, on-demand control of SCI spasticity to greatly improve the quality of life of those affected.

ELIGIBILITY:
Inclusion Criteria:

* SCI adults 18 years and older
* injury levels between C5-T12

Exclusion Criteria:

* severe head injury
* uncontrolled autonomic dysreflexia
* other medical conditions precluding TENS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Ashworth Score | Pre Intervention. 1, 2 and 4 months follow up. In addition, spasticity will be measured every 2 weeks to assess stability of the effects.
  Clinical assessment of spasticity. Scores range from '0' to '4'. Minimum score is '0' meaning no increase in tone. Maximum score is '4' meaning limb is ridged in flexion and extension. The lower the score the better the outcome.

SECONDARY OUTCOMES:
Change in Knee Pendulum Angle | Pre Intervention. 1, 2 and 4 months follow up.
  Clinical assessment of passive knee motion to assess spasticity.
Change in Manual Muscle Testing | Pre Intervention. 1, 2 and 4 months follow up.
  Clinical assessment of muscle strength from grade '0' to '5', where '0' means no strength and '5' means normal strength.
Change in EMG | Pre Intervention. 1, 2 and 4 months follow up.
  Assessment of motor control. Participants are asked to match their muscle contraction force to a target force profile. EMG data will be used to calculate the smoothness of muscle force.
Change in International Standard for Neurological Classification of SCI (ISNCSI) | Pre Intervention. 1, 2 and 4 months follow up.
  Neurological Examination of participant. The Impairment Scale has 5 grades from A to E. Grade A is complete injury and grade E is normal. It is based on the strength of 10 key muscle groups in the upper and lower extremities, sensory response to light touch and pin prick at 28 key sensory points on each side of the whole body, and anal responses.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Gorassini, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta - 524 HMRC, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Only the investigators of this study and the University of Alberta Research Ethics Board will have access to participant information. Only de-identified data will be presented or published.